CLINICAL TRIAL: NCT01304368
Title: Randomized Controlled Pilot Study: Effects of a Heat Pad Application in Patients With Chronic Neck Pain
Brief Title: Effects of Thermotherapy on Chronic Neck Pain
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universität Duisburg-Essen (Other)
Responsible Party: Gustav J Dobos, MD, Universität Duisburg-Essen, Chair of Complementary and Integrative Medicine
Allocation: Randomized | Model: Parallel | Purpose: Treatment
Other Study IDs: 09-3953
Record Dates: First submitted 2011-02-24; First posted 2011-02-25 (Estimated); Last update posted 2011-02-25 (Estimated); Status verified 2011-02

CONDITIONS: Neck Pain
Keywords: Hyperthermia, Induced; Randomized Controlled Trial; Neck Pain; Sensory Thresholds; Pain Measurements
MeSH Terms: conditions — Neck Pain; Hyperthermia | interventions — Hyperthermia, Induced

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Thermotherapy (Active Comparator): Patients are instructed to heat a moor mud filled heat pad (beinio®therm, bb med. product GmbH, Kalkar (Kehrum), Germany) to a hot, but tolerable temperature and to apply it over the painful area once a day for 20 minutes during a period of 14 days. Patients are instructed to continue their usual medication - including analgesic drugs - and physiotherapy (massages and exercise) during the study period.
  Interventions: Procedure: Thermotherapy
- Waiting list (No Intervention): Patients are instructed to continue their usual medication - including analgesic drugs - and physiotherapy (massages and exercise) during the study period.

INTERVENTIONS:
Procedure: Thermotherapy — Patients are instructed to heat a moor mud filled heat pad (beinio®therm, bb med. product GmbH, Kalkar (Kehrum), Germany) to a hot, but tolerable temperature and to apply it over the painful area once a day for 20 minutes during a period of 14 days. Patients are instructed to continue their usual medication - including analgesic drugs - and physiotherapy (massages and exercise) during the study period.
  Arms: Thermotherapy

SUMMARY:
Chronic neck pain is a common worldwide problem. In the majority of cases, patients are treated by medication, referral to a physiotherapist or thermotherapy. Thermotherapy - the therapeutic application of topical heat - provides an easy to apply self-help strategy in patients with chronic neck pain. However, despite the frequent use in clinical practice, there is no research regarding this topic yet.

The aim of this study was to evaluate whether thermotherapy self-treatment for chronic neck pain induces changes in perceived pain intensity and in sensory processing.

ELIGIBILITY:
Inclusion Criteria:

* non-specific neck pain the last 3 months
* mean pain intensity of at least 4 on a 10-level numerical rating scale with "0" meaning "no pain" and "10" meaning "worst pain imaginable"

Exclusion Criteria:

* radicular symptoms
* congenital spine deformity
* skin diseases in the painful area to be treated
* pregnancy
* insulin-dependent diabetes mellitus
* rheumatic diseases
* oncologic diseases
* steroid medication
* anticoagulation medication
* recent invasive or surgical treatment of the spine

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2009-08; Primary Completion 2010-08 (Actual); Study Completion 2010-08 (Actual)

PRIMARY OUTCOMES:
Neck pain intensity (100mm visual analog scale) | Day 14
  100mm visual analog scale

SECONDARY OUTCOMES:
Pain related to motion | Day 14
  100mm visual analog scale for 6 movement directions (flexion, extension, rotation right/left, lateral flexion right/left)
  Reference: Irnich D, Behrens N, Molzen H, König A, Gleditsch J, Krauss M, Natalis M, Senn E, Beyer A, Schöps P. Randomised trial of acupuncture compared with conventional massage and "sham" laser acupuncture for treatment of chronic neck pain. BMJ. 2001 Jun 30;322(7302):1574-8.
Neck disability index (NDI) | Day 14
  The Neck Disability Index is an instrument to assess neck pain complaints.
  Reference: Vernon H, Mior S. The Neck Disability Index: a study of reliability and validity. J Manipulative Physiol Ther 1991;14:409-415.
SF-36 | Day 14
  The SF-36 is a short-form health survey consisting of 8 scales (physical functioning, role-physical, bodily pain, general health, vitality, social functioning, role-emotional, mental health) measuring functional health and well-being as well as a physical a and mental health component scores.
  Reference: Bullinger M, Kirchberger I. SF-36 Fragebogen zum Gesundheitszustand. Göttingen: Hogrefe, 1998.
Pain diary | From day 1 to day 14
  100mm visual analog scale for rating neck pain intensity each day
Pressure pain threshold | Day 14
  Pressure pain threshold measured at two individual points at the neck: (1) at the point of maximal pain and (2) in the adjacent region, one to two cm outside the painful area and at both hands, serving as control sites.
  Measurement procedure according to the protocol of QST.
  Reference: Rolke R et al. Quantitative sensory testing in the German Research Network on Neuropathic Pain (DFNS): standardized protocol and reference values. Pain 2006;123:231-243.
Vibration detection threshold | Day 14
  Vibration detection threshold measured at two individual points at the neck: (1) at the point of maximal pain and (2) in the adjacent region, one to two cm outside the painful area and at both hands, serving as control sites.
  Measurement procedure according to the protocol of QST.
  Reference: Rolke R et al. Quantitative sensory testing in the German Research Network on Neuropathic Pain (DFNS): standardized protocol and reference values. Pain 2006;123:231-243.
Mechanical detection threshold | Day 14
  Mechanical detection threshold measured at two individual points at the neck: (1) at the point of maximal pain and (2) in the adjacent region, one to two cm outside the painful area and at both hands, serving as control sites.
  Measurement procedure according to the protocol of QST.
  Reference: Rolke R et al. Quantitative sensory testing in the German Research Network on Neuropathic Pain (DFNS): standardized protocol and reference values. Pain 2006;123:231-243.
Side effects | Day 14
  Open question on any side effects or other experiences with the treatment
Medication and additional treat ment use | Day 14
  Patient report used medication or additional treatment during the study period

CONTACTS AND LOCATIONS:
Locations (1):
- Kliniken Essen-Mitte, Knappschafts-Krankenhaus, Department for Internal and Integrative Medicine, Essen, North Rhine-Westphalia, Germany